CLINICAL TRIAL: NCT02145325
Title: A Phase I, Single Center Trial of Adoptive Immunotherapy With T-reg Adoptive Cell Transfer (TRACT) to Prevent Rejection in Living Donor Kidney Transplant Recipients
Brief Title: Trial of Adoptive Immunotherapy With TRACT to Prevent Rejection in Living Donor Kidney Transplant Recipients
Acronym: TRACT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Anton Skaro, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00091850
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: End Stage Renal Disease
Keywords: Kidney transplant; Regulatory T cells; Leukopheresis; Immune cells; Stem Cells; Tolerance
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Expanded Tregs (Experimental): Immune cells in the blood will be removed by leukopheresis procedure and stored for later manufacture of subject's Expanded Tregs cellular product. Two months following subject's kidney transplantation, subject will be given an Expanded Tregs infusion intravenously in the Northwestern Clinical Research Unit.
  Interventions: Drug: Expanded Tregs

INTERVENTIONS:
Drug: Expanded Tregs

SUMMARY:
Regulatory CD4+CD25+ T cells (Treg) derived from the thymus and/or peripheral tissues have been demonstrated to broadly control T cell reactivity (14). Importantly, Tregs have been shown to control immune responsiveness to alloantigens and significantly contribute to operational tolerance in transplantation models (15, 16). However, there have been limited efforts to harness the therapeutic potential of directly isolated CD4+CD25+ Treg cells for controlling graft rejection and inducing transplantation tolerance, such as for kidney transplants. In order for CD4+CD25+ Treg cells to be used as a clinical treatment, the following cell properties could be necessary: ex vivo generation of sufficient numbers of cells, migration in vivo to sites of antigenic reactivity, ability to suppress rejection in an alloantigen-specific manner, and survival/expansion after infusion for a critical, but currently unknown, period of time. Our published work and that of other investigators has demonstrated 1) the feasibility of expanding Treg ex vivo, 2) the ability of these cells to downregulate allogeneic immune responses in vitro, and 3) the efficacy of Treg for prevention of allograft rejection in animal models (15,16). We have developed strategies for the ex vivo expansion of naturally occurring human Tregs (nTregs) that allow for the practical employment of this cellular therapy in the clinic. Our central hypothesis is that sufficient human nTreg can be expanded ex vivo and used to both prevent renal transplant rejection and facilitate the reduction and subsequent withdrawal of drug-based immunosuppression. This study will allow for us to define the safety of Treg adoptive cellular transfer (TRACT) in living donor renal transplant recipients that draws upon our extensive preclinical experience with expanded Tregs, as well as our recognized clinical expertise with designing immunosuppressive regimens compatible with this type of therapeutic cell transfer.

DETAILED DESCRIPTION:
Transplantation is the treatment of choice for most causes of end stage renal disease.(1, 2) However, without some modification of the recipient's immune system all allografts succumb to rejection. To prevent this, patients must take immunosuppressive drugs for life, generally a combination of steroids, a calcineurin inhibitor (CNI), such as cyclosporine or tacrolimus, and an antiproliferative agent (azathioprine, mycophenolate mofetil or sirolimus).(3-6) Induction with a brief course of an anti-T lymphocyte antibody preparation (daclizumab, basiliximab, muromonab, alemtuzumab, polyclonal anti-thymocyte globulin) is also used in approximately 70% of U.S. transplant centers.

Dependence on immunosuppression tempers the substantial benefit obtained from transplantation (1-13). The typical regimens are relatively complex and expensive. More importantly, they increase the risk of opportunistic infection and malignancy, and have many non-immune side effects that hamper their tolerability. Specifically, CNIs are nephrotoxic, a side effect of significant concern in renal transplantation. Steroids exacerbate osteoporosis and hyperlipidemia, and cause avascular osteonecrosis. Both classes of agent worsen glucose tolerance and hypertension, and are associated with cosmetic effects causing non-compliance. As such, methods of transplantation that lessen the dependence on chronic immunosuppression stand to reduce the risk and expense of transplantation. They must, however, also prevent rejection. Development of alternate therapies that help to minimize the need for lifelong immunosuppression, or eliminate entirely the need for drugs through the induction of tolerance, are therefore of great interest.

Regulatory CD4+CD25+ T cells (Treg) derived from the thymus and/or peripheral tissues have been demonstrated to broadly control T cell reactivity (14). Importantly, Tregs have been shown to control immune responsiveness to alloantigens and significantly contribute to operational tolerance in transplantation models (15, 16). However, there have been limited efforts to harness the therapeutic potential of directly isolated CD4+CD25+ Treg cells for controlling graft rejection and inducing transplantation tolerance, such as for kidney transplants. In order for CD4+CD25+ Treg cells to be used as a clinical treatment, the following cell properties could be necessary: ex vivo generation of sufficient numbers of cells, migration in vivo to sites of antigenic reactivity, ability to suppress rejection in an alloantigen-specific manner, and survival/expansion after infusion for a critical, but currently unknown, period of time. Our published work and that of other investigators has demonstrated 1) the feasibility of expanding Treg ex vivo, 2) the ability of these cells to downregulate allogeneic immune responses in vitro, and 3) the efficacy of Treg for prevention of allograft rejection in animal models (15,16). We have developed strategies for the ex vivo expansion of naturally occurring human Tregs (nTregs) that allow for the practical employment of this cellular therapy in the clinic. Our central hypothesis is that sufficient human nTreg can be expanded ex vivo and used to both prevent renal transplant rejection and facilitate the reduction and subsequent withdrawal of drug-based immunosuppression. This study will allow for us to define the safety of Treg adoptive cellular transfer (TRACT) in living donor renal transplant recipients that draws upon our extensive preclinical experience with expanded Tregs, as well as our recognized clinical expertise with designing immunosuppressive regimens compatible with this type of therapeutic cell transfer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are males or females age 18-65 years.
2. Donor Age 18-65 years.
3. No prior organ transplant
4. Patients who are single-organ recipients (kidney only).
5. Women who are of childbearing potential must have a negative serum pregnancy test before transplantation and agree to use a medically acceptable method of contraception throughout the treatment period.
6. Subject (recipient) is able to understand the consent form and give written informed consent.

Exclusion Criteria:

1. Known sensitivity or contraindication to sirolimus, tacrolimus or MMF.
2. Patient with significant or active infection.
3. Patients with a positive flow cytometric crossmatch using donor lymphocytes and recipient serum.
4. Patients with PRA >20%
5. Patients with current or historic donor specific antibodies
6. Body Mass Index (BMI) of < 18 or > 35
7. Patients who are pregnant or nursing mothers.
8. Patients whose life expectancy is severely limited by diseases other than renal disease.
9. Ongoing active substance abuse, drug or alcohol.
10. Major ongoing psychiatric illness or recent history of noncompliance.
11. Significant cardiovascular disease (e.g.):

    * Significant non-correctable coronary artery disease;
    * Ejection fraction below 30%;
    * History of recent myocardial infarction.
12. Malignancy within 3 years, excluding nonmelanoma skin cancers.
13. Serologic evidence of infection with HIV or HBVsAg positive.
14. Patients with a screening/baseline total white blood cell count < 4,000/mm3; platelet count < 100,000/mm3; triglyceride > 400 mg/dl; total cholesterol > 300 mg/dl.
15. Investigational drug within 30 days prior to transplant surgery.
16. Anti-T cell therapy within 30 days prior to transplant surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-04; Primary Completion 2016-06-16 (Actual); Study Completion 2016-06-16 (Actual)

PRIMARY OUTCOMES:
Safety Profile Assessment of TRACT | 5 years (60 weeks)
  The primary safety endpoint is the evaluation of cellular related toxicities immediately and within 24 hrs post infusion of TRACT. Since TRACT is being administered to promote immunosuppression and prevent rejection, specific adverse events (subsequent rejection episodes, allosensitization, development of opportunistic infection) within 30 days of infusion will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Skaro, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Comprehensive Transplant Center, Chicago, Illinois, United States